CLINICAL TRIAL: NCT07311278
Title: Identification of Sentinel Lymph Nodes in Breast Cancer Patients Through Non-invasively Fluorescent Imaging Using Indocyanine Green: an International Multicenter Implementation Study.
Brief Title: Identification of Sentinel Lymph Nodes Using Indocyanine Green in Breast Cancer Patients
Acronym: INFLUENCE II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Tessa Dinger, Medical Doctor, St. Antonius Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NL79223.100.22
Record Dates: First submitted 2025-11-26; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: indocyanine green; fluorescence; sentinel lymph node biopsy; sentinel lymph node mapping; sentinel lymph node procedure; ICG; implementation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I: pre-implemtation phase (Other): SLN biopsy using single tracer techentium (current standard)
  Interventions: Procedure: Phase I: Technetium is administered as single tracer to identify the SLN (current standard).
- Phase II: transition phase (Other): SLN biopsy using double tracer technetium and ICG (learning curve)
  Interventions: Procedure: Phase II: SLN biopsy using double tracer technetium and ICG (learning curve)
- Phase III: post-implementation phase (Other): SLN biopsy using single tracer ICG (alternative method)
  Interventions: Procedure: Phase III: ICG is administered as single tracer to identify the SLN (alternative method).

INTERVENTIONS:
Procedure: Phase I: Technetium is administered as single tracer to identify the SLN (current standard). — During this phase, surgeons will use technetium to identify the SLN as this is the current standard of care. This phase will serve as a control group.
  Arms: Phase I: pre-implemtation phase
Procedure: Phase II: SLN biopsy using double tracer technetium and ICG (learning curve) — During this phase, surgeons will primarily use ICG to identify the sentinel lymph node (SLN), while technetium will serve as a control. This approach allows surgeons to gain proficiency with ICG-guided SLN biopsy and safely advance through the learning curve.
  Arms: Phase II: transition phase
Procedure: Phase III: ICG is administered as single tracer to identify the SLN (alternative method). — During this phase, surgeons will use ICG as a singe tracer to identify the SLN.
  Arms: Phase III: post-implementation phase

SUMMARY:
This study aims to evaluate the (inter)national implementation of a new diagnostic method for sentinel lymph node (SLN) detection in breast cancer. While Technetium-99m (99mTc) is the current gold standard for SLN detection, it has drawbacks such as limited availability, logistical challenges, radiation exposure, and potential side effects. Extensive research indicates that Indocyanine Green (ICG) is an equally effective and potentially more practical alternative. Conducting this study will help accelerate the implementation of ICG in clinical practice.

DETAILED DESCRIPTION:
An important part of oncological treatment for breast cancer is determining the lymph node status. A commonly used method for this is the sentinel lymph node (SLN) procedure. Analysis of this node plays a key role in determining both treatment and prognosis.

Currently, the gold standard for SLN localization is the use of Technetium-99m (99mTc). However, this method has several disadvantages. Since not every hospital has a Nuclear Medicine Department, patients often need to be referred to another facility for 99mTc injection and nuclear imaging. This process can be burdensome for patients and poses logistical challenges when scheduling surgeries. In addition, the use of 99mTc involves exposure to radioactive material, and adverse effects such as allergic reactions have been reported. Recent studies have shown that the use of Indocyanine Green (ICG) is equally effective for sentinel lymph node localization as Technetium.

The aim of this study is to evaluate the national and international implementation process of a new diagnostic method for SLN detection.

ELIGIBILITY:
Inclusion Criteria:

* Clinically node-negative, DCIS or invasive breast cancer confirmed by biopsy
* Preoperative axillary ultrasound to confirm clinical node-negative status
* Indication for breast cancer surgery with SLNB via axillar incision
* Written informed consent according to ICH/GCP and national regulations.

Exclusion Criteria:

* Patients < 18 years old.
* Indication for breast cancer surgery with SLNB via mastectomy incision
* Combined MARI procedure
* Known allergy for Indocyanine Green (ICG) or intravenous contrast or iodine
* History of axillary lymph node dissection
* Hyperthyroidism or thyroid cancer
* Pregnancy or breast-feeding
* Psychological, familial, sociological or geographical factors that could potentially hamper compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Identifaction rate | Perioperatively
  Identification rate is defined as the proportion of patients in whom lymph nodes were identified with the gamma-probe using technetium or the fluorescent signal of ICG.

SECONDARY OUTCOMES:
Number of lymph nodes identified | Perioperatively
  This indicates the total number of lymph nodes identified with ICG or technetium.
Percentage of SLNs identified per tracer | Perioperatively
  Percentage of SLNs that had technetium uptake / were fluorescent.
Pathology assesment per SLN | Perioperatively
  The pathology of the identified SLN during surgery
Detection time | Intraoperatively
  Time in minutes to excise the SLN, measured from start of SLN procedure until detection of the first SLN.
Complications | From the time of the SLN procedure up until three weeks of follow-up.
  Complications including (wound)infection, bleeding, seroma, and mild allergic reaction.
Adverse events | Monitored during study period until one year of follow-up
  Number of adverse events attributable to technetium or ICG.
Locoregional recurrence at 1 year follow-up | Until the end of the study (after 1 year of follow-up)
Surgeon's expectations regarding ICG | Pre-implementation (prior to the transion phase)
  Expectations of the participating surgeons regarding the use of ICG for SLN procedure using a study-specific survey with open-ended questions and multiple choice items.
Surgeons' experiences regarding ICG | Up to 12 months after transition to ICG as single tracer
  Experiences of the participating surgeons regarding the use of ICG for SLN procedure using a study-specific survey with open-ended questions and multiple choice items.
Learning curve per surgeon | From each surgeon's first procedure using the double tracer method (technetium and ICG) through completion of the transition phase, assessed over up to 12 months.
  The learning curve process will be expressed by visualizing inter-surgeon variability in the number of procedures required to achieve proficiency portrayed in a scatterplot.

CONTACTS AND LOCATIONS:
Locations (11):
- Ospedale Pederzoli, Peschiera del Garda, Italy
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - FlevoZiekenhuis, Almere Stad
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - HagaZiekenhuis, The Hague
  - Bernhoven Ziekenhuis, Uden
  - Isala Ziekenhuis, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided